CLINICAL TRIAL: NCT05811507
Title: Evaluation of Serum Adrenal Androgens Among Prepubertal and Pubertal Boys With Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salma Samir Ismail, assistant lecturer of pediatrics, Sohag University
Other Study IDs: Soh-Med-23-03-03MD
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases group of patients:: It will include patients with autism spectrum disorder..
  Interventions: Diagnostic Test: serum total testosterone, serum androsterone, serum androstenedione and serum dehydroepiandrosterone sulfate; Diagnostic Test: The Childhood Autism Rating Scale (CARS); Diagnostic Test: DSM-5 Diagnostic Criteria for ASD; Diagnostic Test: Assesment of IQ: The Stanford-Binet V (Stanford-Binet Intelligence Scales):
- control group of patients:: It will include healthy boys who don't have any manifestations of ASD according to DSM-V Criteria and CARS score, and are age and Tanner stage matched to cases.
  Interventions: Diagnostic Test: serum total testosterone, serum androsterone, serum androstenedione and serum dehydroepiandrosterone sulfate; Diagnostic Test: The Childhood Autism Rating Scale (CARS); Diagnostic Test: DSM-5 Diagnostic Criteria for ASD; Diagnostic Test: Assesment of IQ: The Stanford-Binet V (Stanford-Binet Intelligence Scales):

INTERVENTIONS:
Diagnostic Test: serum total testosterone, serum androsterone, serum androstenedione and serum dehydroepiandrosterone sulfate — Venous blood samples will be collected into sterile EDTA tubes around 10 am. Blood taken from controls will be collected at the same time. All samples will be delivered into the laboratory immediately after collection and centrifuged at 3000 × g, 4 °C for 10 min. Plasma samples were stored at -80 °C until the analysis using ELIZA
Diagnostic Test: The Childhood Autism Rating Scale (CARS) — It is done by rating the child's behaviors from 1 to 4. 1 being normal for your child's age, 2 for mildly abnormal, 3 for moderately abnormal, and 4 as severely abnormal. Scores range from 15 to 60 with 30 being the cutoff rate for a diagnosis of mild autism. Scores 30-37 indicate mild to moderate autism, while scores between 38 and 60 are characterized as severe autism
Diagnostic Test: DSM-5 Diagnostic Criteria for ASD — Persistent deficits in social communication and social interaction across multiple contexts. Restricted, repetitive patterns of behavior, interests, or activities. Symptoms must be present in the early developmental period, Symptoms cause clinically significant impairment in social, occupational, or other important areas of current functioning.These disturbances are not better explained by intellectual disability or global developmental delay.
Diagnostic Test: Assesment of IQ: The Stanford-Binet V (Stanford-Binet Intelligence Scales): — IQ Score ranges for the Stanford-Binet:
  Low average: 80-89 Average: 90-109 High average: 110-119 High achiever: 120-129 Moderately gifted: 130-144 Highly gifted: 145-160+

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder of unclear etiology. There are theories depicting the importance of sex steroid hormones in autism, since the prevalence of the disorder is male-biased. What makes boys more vulnerable to achieve the diagnosis of autism remains unclear. One of the theories strengthens the importance of fetal organizational effect of testosterone on brain development. Baron Cohen with coworkers showed that elevated fetal levels of several androgens including testosterone were high in male-fetuses who later in postnatal life achieved the diagnosis of autism and fetal testosterone levels were positively correlated with autistic traits in general population.

Females with conditions of abnormal prenatal exposure to testosterone and its sex steroid precursors, such as congenital adrenal hyperplasia and polycystic ovary syndrome, were found to have higher rate of autistic traits as well as their children were of higher risk of developing autism. However, the exact mechanism by which these hormones influence the manifestation of autistic traits remains undiscovered. Another model explaining higher prevalence of ASD in males is a female protective model which suggests that multiple genetic factors contribute to the development of ASD and that higher threshold of genetic liability is required in females compared to males. Zhang et al. demonstrated genetic evidence of sex differences in ASD confirming female protective model, employing investigation of de novo mutations, common variants of ASD candidate genes and their co-expression in male and female brain.

During infancy: The Gonadotropin releasing hormone (GnRH) pulse generator is reactivated by 6 to 10 days after birth. This period, termed the mini puberty of infancy, was first described in the 1970s. During mini puberty, luteinizing hormone (LH) levels approximate pubertal concentrations, reaching a peak between 16 and 20 days of life. Serum testosterone levels rise in response to rising concentrations of LH, paralleling an increase in Leydig cell number and testicular testosterone concentrations. Serum testosterone levels peak from 1 to 3 months (210 ± 130 ng/dL or 7.28 ± 4.51 nmol/L on day of life 30) and decline by roughly 50% per month reaching prepubertal levels by 7 to 12 months of age. Dihydrotestosterone (DHT) concentrations parallel the rise in testosterone, reaching pubertal values during the early postnatal period.

During puberty: Testosterone is produced primarily by the testes, though a small amount is also made in the adrenal gland. Gonadarche refers to the onset of sex steroid production from the gonads and occurs in response to pulsatile production of GnRH from the hypothalamus, which in turn stimulates production of LH and Follicle stimulating hormone (FSH) from the pituitary gland. LH stimulates the Leydig cells to produce testosterone, whereas FSH stimulates the Sertoli cells to proliferate and initiate spermatogenesis.

Active androgens are synthesized via two alternative pathways. The first of them is known as the classic "frontdoor" pathway with pregnenolone serving as androgen precursor, which underwent a conversion to DHEA and subsequently to androstenediol. These metabolic steps are catalyzed by CYP17A1 (in the C17,20-lyase step) and (mostly adrenal) AKR1C3 enzyme, respectively. Dehydroepiandrosterone (DHEA) and androstenediol are readily sulfated by SULT2A1 in adrenal cortex and their sulfates serve as the stock pool for the production of active androgens of the adrenal origin as the production of androgens in early childhood of boys is limited to extra-gonadal tissues, such as adrenal, skin, etc. These sulfated primary androgens may be subsequently deconjugated and metabolized by HSD3B1 and HSD3B2 isoforms to androstenedione and Total testosterone (TST) and then to 5α/β-reduced 17-oxo- and 17β-androgens, respectively. In addition, the androstenedione may be readily converted to testosterone by adrenal AKR1C3. From the aforementioned substances, TST, 5α-dihydrotestosterone, and 11-oxo-testosterone are known as the most potent bioactive androgens. Besides the "frontdoor" pathway the dihydrotestosterone may be also formed by so called "backdoor" pathway. This pathway is based on a direct conversion of 5α/β-reduced pregnane steroids (C21) to their 5α/β-reduced androgen (C19) metabolites which is catalyzed by the same enzyme converting pregnenolone to DHEA (CYP17A1 in the C17,20-lyase step). These 5α/β-reduced androgen (C19) metabolites include also the most active androgen 5α-dihydrotestosterone. The "backdoor" pathway is crucial for androgen synthesis in marsupials but may also be active in various human steroid-related disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-18 years
2. Proved diagnosis by clinical manifestations of ASD in addition to DSM-V Criteria
3. Assessment of ASD severity by Childhood Autism Rating Scale (CARS)

Exclusion Criteria:

1. Those with history of metabolic and neurodegenerative disease
2. Medication History: Those on long-term use of antibiotics, non-steroidal drugs, immune-stimulants or immune-suppressive drugs
3. Those with structural brain abnormalities
4. Those with audiological or visual problems
5. Those with other psychiatric problems
6. Those with history of systemic illness as allergic disease, immunodeficiency or autoimmune disease

Ages: 6 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Age: 6-18 years. Proved diagnosis by clinical manifestations of ASD in addition to DSM-V Criteria. Assessment of ASD severity by Childhood Autism Rating Scale (CARS)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
serum total testosterone level. | baseline
  serum total testosterone level will be measured in (nglml).
serum dehydroepiandrosterone sulfate (DHEAS) level | baseline
  serum dehydroepiandrosterone sulfate (DHEAS) will be measured in (mcgldl)
serum androsterone level | baseline
  serum androsterone level will be measured in (nglml)
serum androstenedione level | baseline
  serum androstenedione level will be measured in (nglml)
Assessment of severity of autism | baseline
  Assessment of severity of autism by Childhood Autism Rating Scale (CARS)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Baron-Cohen S, Auyeung B, Norgaard-Pedersen B, Hougaard DM, Abdallah MW, Melgaard L, Cohen AS, Chakrabarti B, Ruta L, Lombardo MV. Elevated fetal steroidogenic activity in autism. Mol Psychiatry. 2015 Mar;20(3):369-76. doi: 10.1038/mp.2014.48. Epub 2014 Jun 3. PMID 24888361
- [Background] Cherskov A, Pohl A, Allison C, Zhang H, Payne RA, Baron-Cohen S. Polycystic ovary syndrome and autism: A test of the prenatal sex steroid theory. Transl Psychiatry. 2018 Aug 1;8(1):136. doi: 10.1038/s41398-018-0186-7. PMID 30065244
- [Background] Robinson EB, Lichtenstein P, Anckarsater H, Happe F, Ronald A. Examining and interpreting the female protective effect against autistic behavior. Proc Natl Acad Sci U S A. 2013 Mar 26;110(13):5258-62. doi: 10.1073/pnas.1211070110. Epub 2013 Feb 19. PMID 23431162
- [Background] Zhang Y, Li N, Li C, Zhang Z, Teng H, Wang Y, Zhao T, Shi L, Zhang K, Xia K, Li J, Sun Z. Genetic evidence of gender difference in autism spectrum disorder supports the female-protective effect. Transl Psychiatry. 2020 Jan 15;10(1):4. doi: 10.1038/s41398-020-0699-8. PMID 32066658